CLINICAL TRIAL: NCT04560543
Title: Prophylactic Laparoscopic Suspension After McCall - Benefit and Longterm Outcome
Brief Title: Prophylactic Laparoscopic Suspension After McCall
Acronym: LAPCALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-01046
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Prolapse Pelvic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McCall suture (Experimental): Uterus removal by laparoscopy with usual vaginal closure and additional (McCall) suture, which is intended to prevent descent.
  Interventions: Procedure: McCall suture
- standard cuff closure (Sham Comparator): Uterus removal by laparoscopy with usual vaginal closure without additional (McCall) suture. (as performed so far)
  Interventions: Procedure: Standard cuff closure

INTERVENTIONS:
Procedure: McCall suture — Laparoscopic suture including the uterosacral ligaments and the peritoneum
  Other Names: Uterosacral Ligament Suspension
  Arms: McCall suture
Procedure: Standard cuff closure — Standard laparoscopic barbed suture of the vaginal cuff
  Arms: standard cuff closure

SUMMARY:
There is prove of prolapse prevention in vaginal hysterectomy using the McCall suture. Poor and especially no long-term data exists for a standardized laparoscopic approach, but the few studies could show good anatomic results.

The aim is to test the effectiveness of the laparoscopic McCall suture compared to usual vaginal cuff closure in a randomized controlled double-blinded trial.

DETAILED DESCRIPTION:
182 patients will be enrolled in the study. We randomize the patient before surgery and information about the procedure will be transmitted to the theatre in a sealed envelope. The surgeon will open the envelope just before surgery. For randomization we apply a 1:1 allocation (standard vaginal cuff closure VS standard vaginal cuff closure with McCall sutures). The McCall suture is standardized: we apply a purse-string suture including both USL and the peritoneum.

Follow-up visits measuring POP-Q are planned after 6 weeks and yearly until 5 years.

ELIGIBILITY:
Inclusion criteria

* LSC simple hysterectomy,
* Neg. SS test if premenopausal
* >18j,
* Consent to participate in the study
* Understanding of the German language

Exclusion criteria

* Prolapse as indication for surgery
* Known or suspected non-compliance
* Additional incontinence procedures
* Patients with deep infiltrating endometriosis
* Irradiation pre- or postoperative
* Pregnancy and lactation.
* Transgender population
* Conversion from laparoscopy to laparotomy
* Inability to understand the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 182 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Prolapse of the apical compartment. Primary Quantification by the Pelvic organ prolapse Scoring system (POP-Q) Depending on vaginal length, it could vary between +10 and -10cm. | 5 years
  Primary Quantification by the Pelvic organ prolapse Scoring system (POP-Q), ranges from -10 (low) to +10 (high), better outcome with higher score endpoint is the prolapse of the apical compartment (point D in the POP-Q score, vaginal dome in relation to the hymen) after 5 years.
  Point D is a value measured in centimeters. Depending on vaginal length, it could vary between +10 and -10cm. Reference point of all measurements is the hymen.

SECONDARY OUTCOMES:
Sexual function | 5 years
  Quantification by the Female Sexual Function Index, Score 0 - 5, better outcome with higher score

CONTACTS AND LOCATIONS:
Overall Officials: Michel D Mueller, Prof., Study Director — Department of Gynaecology, University Hospital, Berne
Locations (1):
- Universitätsfrauenklink Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No